CLINICAL TRIAL: NCT03086525
Title: The Influence of Beliefs (Fear of Movement, Pain-related Fear, Self-efficacy, and Pain Acceptance) in the Development and/or Perpetuation of Muasculoskeletal Pain. Protocol
Brief Title: Influence of Beliefs on the Development of Musculoskeletal Pain.
Status: Completed | Type: Observational
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Other Study IDs: UNOMalaga
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2019-12

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic pain; Psychological factors; Musculoskeletal pain; Prognosis
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Musculoskeletal pain: Participants Healthy male and female students, students of the University of Málaga, will be recruited. . The inclusion criteria are as follows: (i) men / women over 18 years; (ii) students of the University of Málaga.
  Interventions: Other: Diagnosis/Prognosis

INTERVENTIONS:
Other: Diagnosis/Prognosis — The present study will be a prospective observational study of 4 years that will be carried out between September 2017 and September 2020 at the University of Malaga. Several questionnaires assessing different beliefs associated with pain will be administered to participants. The results will be evaluated at baseline (t1) and in 4 follow-ups (at 12 (t2), 24 (t3), 36 (t4) and 48 (t5) months.

SUMMARY:
Musculoskeletal pain is highly prevalent, disabling, and with high socio-economic costs, with many negative effects on quality of life. It affects the ability to perform work, social, recreational and domestic tasks, changing the mood and concentration of this population. Despite the worldwide prevalence and socioeconomic burden of this condition, a clear understanding of its etiology and pathogenesis remains elusive.

Aims:

(i) to analyze the possible level of association between fear of pain, fear of movement, self-efficacy, and pain acceptance on pain-disability at the start of the study and prospectively evaluate its role as a risk factor; (ii) to evaluate the possible role as a prognostic factor of fear of pain, fear of movement, self-efficacy and pain acceptance in those who develop musculoskeletal pain at follow-up; (iii) explore the possible mediating power of fear of movement and self-efficacy in the relationship between pain-disability; (iv) investigate what percentage of the variance accounts for beliefs (fear of pain, fear of movement, self-efficacy, and acceptance of pain) in predicting the onset and / or maintenance of musculoskeletal pain.

DETAILED DESCRIPTION:
The present study will be a prospective observational study of 4 years that will be carried out between September 2017 and September 2020 at the University of Malaga. Several questionnaires assessing different beliefs associated with pain will be administered to participants. The results will be evaluated at baseline (t1) and in 4 follow-ups (at 12 (t2), 24 (t3), 36 (t4) and 48 (t5) months. It will be implemented and reported in line with the SPIRIT statement and the STROBE guidance.

Participants A consecutive sample of healthy male and female students, students of the University of Málaga, will be recruited. Research assistants trained by the principal investigator will be in charge of carrying out the recruitment and evaluating the participants for their eligibility. Participants who meet the inclusion criteria will be invited to participate in this study, and then evaluated at baseline and at 12, 24, 36 and 48 months of follow-up. The inclusion criteria are as follows: (i) men / women over 18 years; (ii) students of the University of Málaga belonging to one of the disciplines previously mentioned. The exclusion criteria are as follows: (i) participants currently experiencing musculoskeletal pain; (ii) participants currently taking medication; (iii) previous histories of musculoskeletal surgery; (Iv) inability to provide written informed consent and / or complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* men / women over 18 years.
* students of the University of Málaga.

Exclusion Criteria:

* participants currently experiencing musculoskeletal pain.
* participants currently taking medication.
* previous histories of musculoskeletal surgery.
* inability to provide written informed consent and / or complete questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects between 18-80 years without musculoskeletal pain, and students of the university of malaga
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline the numerical pain rating scale (NRS) at 12,24,36,48 months | Pain will be evaluated at baseline and 4 follow-ups (12.24.36.48 months).
  Pain: The Numerical Rating Scale (NRS) will assess the pain intensity of each patient at baseline and prospectively. NRS scores range from 0 to 10, with 0 without pain and 10 with the worst pain imaginable. It has been shown that the NRS has a good test-retest reliability of the same day.

SECONDARY OUTCOMES:
Change from baseline the pain disability questionnaire (PDQ) at 12,24,36,48 months | Disability will be evaluated at baseline and 4 follow-ups (12,24,36,48 months)
  The Pain Disability Questionnaire (PDQ) is a 15-question questionnaire that evaluates musculoskeletal disorders focusing on disability and the ability of patients to perform activities of daily living. The marker ranges from 0 (optimal function) to 150 (total disability).

OTHER OUTCOMES:
Change from baseline the tampa scale for kinsiophobia (TSK-11) at 12,24,36,48 months | Fear of movement will be evaluated at baseline and 4 follow-ups (12,24,36,48 months)
  Fear of movement: The short version of the Tampa Scale for Kinesiophobia (TSK-11) will be used to assess fear of movement
Change from baseline the fear pain questionnaire (FPQ-III) at 12,24,36,48 months | Pain-related fear will be evaluated at baseline and 4 follow-ups (12,24,36,48 months)
  Pain-related fear: The short version (9-items) of the Fear of Pain Questionnaire (FPQ-III) will be used to assess the fear of pain in this population
Change from baseline the chronic pain acceptance questionnaire (CPAQ) at 12,24,36,48 months | Pain acceptance will be evaluated at baseline and 4 follow-ups (12,24,36,48 months)
  Pain acceptance: The Chronic Pain Acceptance Questionnaire (CPAQ) will measure pain acceptance through 20 items
Change from baseline the pain self-efficacy questionnaire (PSEQ) at 12,24,36,48 months | Self-efficacy will be evaluated at baseline and 4 follow-ups (12,24,36,48 months)
  Self-efficacy: The Pain Self-Efficacy Questionnaire (PSEQ) contains 10 questions that will measure the patient's confidence in performing certain activities despite pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga
Locations (1):
- Univeristy of Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No